CLINICAL TRIAL: NCT06762470
Title: Prognostic Value of Pretreatment Peripheral Circulating Lymphocyte CD4/CD8 Ratio in Patients with Non-metastatic Nasopharyngeal Carcinoma: a Multi-center Prospective Observational Study
Brief Title: Prognostic Value of CD4/CD8 Ratio in Patients with Nasopharyngeal Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKJP1320242038
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Histopathological Diagnosis of Nasopharyngeal Carcinoma; Patients with Nasopharyngeal Carcinoma Without Distant Metastases After AJCC/UACC 8th Edition
Keywords: nasopharyngeal carcinoma; Peripheral blood circulating lymphocytes before treatment; CD4/CD8 ratio; Prognostic value
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High CD4/CD8 ratio group: High CD4/CD8 ratio of peripheral blood lymphocytes before treatment: CD4/CD8 ratio ≥1
- Low CD4/CD8 ratio group: Low CD4/CD8 ratio of peripheral blood lymphocytes before treatment: CD4/CD8 ratio <1

SUMMARY:
In our previous retrospective study, we identified circulating immune cell counts and the CD4/CD8 ratio as significant prognostic markers in nasopharyngeal carcinoma. Building on these findings, this study aims to conduct a multi-center prospective observational study to evaluate the prognostic value of the circulating lymphocyte CD4/CD8 ratio in nasopharyngeal carcinoma patients prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histopathological diagnosis of nasopharyngeal carcinoma;2.Patients with nasopharyngeal carcinoma without distant metastases after AJCC/UACC 8th edition;3.The radiation therapy technique is IMRT;4.Age 18-70 years;5.Has good organ function;6.Patients who are willing and able to comply with visit schedules, treatment plans, laboratory tests, and other study procedures; 7.Willing to comply with the arrangement during the study period and can no longer participate in any other clinical studies related to drugs and medical devices;8.Patients sign a formal informed consent form to indicate that they understand that this study is in accordance with the hospital's policies.

Exclusion Criteria:

* 1.Concomitant with other tumors;2.Those with a history of severe immediate allergies to any of the drugs used in this study;3.Lack of or limited capacity for civil conduct;4.Addiction to drugs or alcohol, with a physical or psychiatric disorder;5.Previous diagnosis of immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related disease;6.Pregnant or lactating female patients, male or female patients of childbearing potential who are unwilling or unable to use contraception throughout the study period and for at least 1 year after the end of the treatment regimen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 Years
  The time from the first diagnosis of nasopharyngeal carcinoma to the first observation of disease progression or death from any cause

SECONDARY OUTCOMES:
Overall Survival | 3 Years
  The time from the first diagnosis of nasopharyngeal carcinoma to the occurrence of death from any cause
Distant Metastasis-free Survival | 3 years
  Distant metastasis-free survival (DMFS) was defined as the time from diagnosis to the occurrence of distant metastasis or the date of censoring, whichever came first.
Locoregional Recurrenc-free Survival | 3 Years
  Locoregional recurrence-free survival (LRRFS) was defined as the time from diagnosis to the occurrence of locoregional recurrence or the date of censoring, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tao CJ, Chen YY, Jiang F, Feng XL, Jin QF, Jin T, Piao YF, Chen XZ. A prognostic model combining CD4/CD8 ratio and N stage predicts the risk of distant metastasis for patients with nasopharyngeal carcinoma treated by intensity modulated radiotherapy. Oncotarget. 2016 Jul 19;7(29):46653-46661. doi: 10.18632/oncotarget.9695. PMID 27270307
- [Background] Gu Y, Jin Y, Ding J, Yujie W, Shi Q, Qu X, Zhao S, Li J, Lijuan C. Low absolute CD4+ T cell counts in peripheral blood predict poor prognosis in patients with newly diagnosed multiple myeloma. Leuk Lymphoma. 2020 Aug;61(8):1869-1876. doi: 10.1080/10428194.2020.1751840. Epub 2020 Apr 23. PMID 32324088